CLINICAL TRIAL: NCT06572761
Title: A Combination of Antibiotics to Decrease Neonatal Mortality and Morbidity for Pregnancies Complicated With Previable Labour and Intact Membranes: a Multicenter, Open-label, Randomized and Controlled Trial
Brief Title: A Combination of Antibiotics to Decrease Neonatal Morbidity and Mortality for Previable Threatened Labor
Acronym: ECHEC-MAT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP220670; 2023-505500-37-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Previable Labour With Intact Membranes
Keywords: previable labour; preterm
MeSH Terms: conditions — Premature Birth | interventions — Ceftriaxone; Clarithromycin; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination of antibiotics (Experimental): Combination of antibiotics (3rd generation of cephalosporin, clarithromycin, metronidazole)
  + routine care (emergency cerclage, vaginal progesterone)
  Interventions: Drug: Combination of antibiotics; Device: Emergency cerclage; Drug: Vaginal progesterone
- Routine care (Active Comparator): Routine care (emergency cerclage, vaginal progesterone)
  Interventions: Device: Emergency cerclage; Drug: Vaginal progesterone

INTERVENTIONS:
Drug: Combination of antibiotics — Ceftriaxone : 1g/day parenteral clarithromycin 500 mg*2/day orally metronidazole 500mg*3/ day orally
  Other Names: Ceftriaxone; clarithromycin, metronidazole
  Arms: Combination of antibiotics
Device: Emergency cerclage — Emergency cerclage
Drug: Vaginal progesterone — Vaginal progesterone

SUMMARY:
The purpose of this study is to determine whether a combination of antibiotics (cephalosporin 3rd generation, clarithromycin, metronidazole) are effective to prolong pregnancies complicated with previable threatened labour with intact membranes.

DETAILED DESCRIPTION:
Observational data suggest that subclinical infectious conditions can lead to spontaneous preterm labor. 10% of births are premature, but the morbidity/mortality of premature babies is concentrated mainly among newborns born before 30 weeks of gestation or weighing less than 1500 g. The relationship to infection/inflammation and premature birth is not constant throughout pregnancy, but this infectious risk increases the earlier the gestational age of spontaneous labor is (before 30 weeks). The pathogens that have the strongest associations with premature birth are Gardnerella vaginalis, Ureaplasma urealyticum and Mycoplasma hominis, but also Streptococcus B, Escherichia coli, Klebsiella spp, or Haemophilus influenzae.

Antibiotic treatment to treat an intra-amniotic infection is considered ineffective. Indeed, the last randomized trial (Oracle 2, 2001), which studied several antibiotic regimens for threatened premature delivery with intact membranes, did not find a significant reduction in neonatal morbidity/mortality after administration of co-beta-lactam, erythromycin or the combination of both. In addition, this large trial dominates the results of the latest Cochrane meta-analysis which evaluated preventive antibiotic therapy to stop premature labor with intact membranes.

Recently, it has been showed that a new combination of antibiotics (ceftriaxone, clarithromycin and metronidazole) reduced the risk of infection and intra-amniotic inflammation in preterm labor with intact membranes. This retrospective study deserves to be confirmed by a randomized study

The investigator's goal is to study whether a new combination of antibiotics in a very limited population of pregnancies complicated by the threat of late miscarriage would make it possible to prolong pregnancies in order to improve neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Threatened previable prelabor with intact membranes between 18weeks of gestation +0/7 and 23 weeks of gestation 6/7 SA defined on endovaginal ultrasound by a short cervix ≤10 mm, and/or protrusion of the membranes on speculum examination.
* Maternal age >18 years
* Affiliated with social security
* Correct understanding of the French language
* Singleton pregnancy
* Foetus alive at time of inclusion
* Absence of regular and painful uterine contractions

Exclusion Criteria:

* Premature labor defined by regular, painful uterine contractions and a short cervix
* Protected person (patient under guardianship/curatorship/or legal protection)
* Multiple pregnancies
* Premature rupture of membranes
* Acute chorioamnionitis
* Contraindication to protocol antibiotics
* Chromosomal abnormality, congenital malformation
* Patients who received antibiotics before randomization, or requiring antibiotics for another indication (chorioamnionitis, pyelonephritis, etc.)
* Participation in another research (Specify the category: RIPH, EC, IC, etc.) or being in the exclusion period following previous research involving humans, if applicable
* Patient under AME (if no exemption from affiliation)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
A perinatal composite outcome | Up to 24 weeks
  * Late miscarriage
  * Perinatal mortality
  * Bronchodysplasia,
  * Sepsis proven by blood culture,
  * Intraventricular hemorrhage ≥3,
  * Periventricular leukomalacia ≥2,
  * Ulcero-necrotizing enterocolitis at stage ≥2 according to the Bell classification.

SECONDARY OUTCOMES:
Gestationnal age at delivery | 6 months
  * Gestationnal age at delivery ≥ 24 weeks of gestation (wg) 0/7, 28 wg0/7, 32 wg0/7, 34 wg0/7 et 37 wg0/7
  * Latency period between randomisation and delivery (≥2 days, ≥7 days, ≥14 days et ≥28 days)
Maternal Morbidty | 6 months
  Chorioamniotitis, postpartum endometritis , sepsis proven par positive hemocultures
Bacteriological | 6 months
  Acquisition of multi-resistant germs during childbirth

CONTACTS AND LOCATIONS:
Overall Officials: Thibaud QUIBEL, MD, PhD, Principal Investigator — Centre Hospitalier Poissy-Saint Germain; Jean BOUYER, Study Chair — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Centre Hospitalier Poissy-Saint Germain, Poissy, France